CLINICAL TRIAL: NCT03084406
Title: Web-Based Tool for the Dissemination of Evidence-based Interventions for ATOD
Brief Title: Efficacy of Centervention-ATOD: An Implementation Tool for Dissemination of Evidence-based Programs for Substance Abuse
Acronym: CV-ATOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 3-C Institute for Social Development (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R44DA035014 (NIH)
Record Dates: First submitted 2017-03-02; First posted 2017-03-21 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Substance Abuse
Keywords: Substance Abuse; Implementation Science; Evidence-based Practices
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: The pilot test will employ a Hybrid Type II study design to simultaneously test the clinical evidence-based program as well as the implementation strategy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Implementation (EI) (Experimental): Providers in the Free Talk EI condition will receive access to CV-ATOD. They will participate in an online training course that mirrors the training in the IAU condition. EI providers will also receive access to interactive online exercises and practice activities within the training module. They will have online access to the Free Talk: Group MI for Teens searchable manual and materials via CV-ATOD. Providers may complete an optional CE course following the completion of the training module. EI providers will have access to all EBP implementation tools provided by CV-ATOD. Student providers in the CHOICE EI condition will receive access to CV-ATOD. They will participate in an online training course that mirrors the training in the IAU condition. However, EI providers will also receive access to interactive online exercises and practice activities within the training module. They will have online access to the CHOICE: Group MI for Teens searchable manual and materials via CV-ATOD.
  Interventions: Other: Centervention-ATOD (CV-ATOD)
- Implementation As Usual (IAU) (No Intervention): CMH providers in the Free Talk IAU condition will receive access to the Group MI for Teens website that provides asynchronous, self-paced training videos as well as downloadable intervention materials and resources. CMH providers in this condition are only required to watch the first two training videos before receiving access to download the Free Talk training manual and materials. Providers may also complete an optional CE course following the completion of all training videos. Student providers in the CHOICE IAU condition will receive access to the Group MI for Teens website that provides online training videos as well as downloadable intervention materials and resources. IAU providers are only required to watch the first two training videos before receiving access to download the CHOICE training manual and materials. Providers may also complete an optional EBP knowledge test following the completion of all training videos.

INTERVENTIONS:
Other: Centervention-ATOD (CV-ATOD) — A customizable suite of online tools specifically designed to support quality implementation and sustainability of any ATOD-EBP within real-world service settings.
  Arms: Enhanced Implementation (EI)

SUMMARY:
The pilot test of Centervention-ATOD, a customizable suite of online tools specifically designed to support quality implementation and sustainability of any ATOD-EBP within real-world service settings, will evaluate whether the product awards additive benefits in provider implementation proficiency and efficacy, quality of implementation delivery, and EBP (i.e., Free Talk or CHOICE) outcomes compared to traditional implementation methods. Additionally, a cost-effectiveness study will be conducted to assess whether the implementation support strategy (i.e., Centervention-ATOD) is more cost-effective than traditional implementation methods.

DETAILED DESCRIPTION:
Alcohol, tobacco, and other drug (ATOD) use among adolescents is a major public health problem with devastating personal, familial, and societal costs. Substance use in youth is associated with increased accidental injuries (including overdoses), psychiatric comorbidities, suicidality, school problems, juvenile delinquency, social and family problems, sexual impulsivity, and health consequences.A burgeoning neuroscience literature demonstrates ATOD use in youth is associated with a host of negative and potentially long-term sequelae, including alterations in brain structure, function, and neurocognition. Moreover, drug use in adolescence is the best predictor of abuse in adulthood; data published by the National Center on Addiction and Substance Abuse reveal that 90% of adults who meet substance dependence criteria began using alcohol and drugs during adolescence. In the U.S., the economic impact of substance abuse is staggering: in 2005, federal, state, and local governments spent a combined $467 billion on the direct and indirect costs associated with addiction, rendering substance dependence the largest, costliest, and most preventable public health problem in the U.S. today.

Over the past few decades, significant progress has been made in the field of ATOD research in developing evidence-based practices (EBPs), with research demonstrating ATOD users who receive research-proven treatments are nearly 2.5 times more likely to achieve clinically significant post-treatment abstinence compared to those receiving non-evidence-based treatment. However, despite availability, EBPs are rarely adopted for use in everyday service settings. Further, even when adopted, considerable variation exists both in the quality with which EBPs are implemented and their long-term sustainability. Furthering our understanding of how efficacious treatment programs can be successfully introduced into real-world treatment settings is key to bridging this research-to-practice gap.

The pilot test of Centervention-ATOD, a customizable suite of online tools specifically designed to support quality implementation and sustainability of any ATOD-EBP within real-world service settings, will evaluate whether the product awards additive benefits in provider implementation proficiency and efficacy, quality of implementation delivery, and EBP (i.e., Free Talk or CHOICE) outcomes compared to traditional implementation methods. Additionally, a cost-effectiveness study will be conducted to assess whether the implementation support strategy (i.e., Centervention-ATOD) is more cost-effective than traditional implementation methods.

The pilot test will employ a Hybrid Type II study design[14] to simultaneously test the clinical evidence-based program as well as the implementation strategy. Regardless of the EBP implemented, 110 mental health (MH) providers will be randomly assigned to one of two conditions: (1) Enhanced implementation (EI) or (2) Implementation as Usual (IAU). Providers will either implement (a) Free Talk, a motivational interviewing group intervention with 5-8 youth per group over a six-week period or (b) CHOICE, a motivational interviewing group prevention program with 5-8 youth per group over a five-week period. Participating youth between ages 14-17 who may have experimented with alcohol or other drugs (AOD) will participate in the Free Talk intervention while youth between ages 11-15 who may or may not have used any substances will participate in the CHOICE prevention program. At the conclusion of the pilot test, a study of cost-effectiveness of the implementation support strategy (i.e., Centervention-ATOD) will be conducted with agency administrators of participating providers.

ELIGIBILITY:
Inclusion Criteria: Community Mental Health (CMH) Providers

* Licensed CMH Provider to youth between ages 14 -17 for Free Talk EI/TAU
* Students enrolled in local University Clinical Programs for CHOICE EI/TAU

Inclusion Criteria: Youth

* Between ages 14 -17 for Free Talk EI/TAU, Between ages 11 -14 for CHOICE EI/TAU
* For Free Talk EI/TAU, youth may have experimented with or currently use alcohol or other drugs.
* For CHOICE EI/TAU, youth may, or may not, have considered ATOD experimentation.

Ages: 11 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2017-12-22 (Actual)

PRIMARY OUTCOMES:
Change in Provider EBP knowledge and MI skills | 1) prior to starting the trial (baseline) but after completing the training for the EBP and the ISS 2) within two weeks of completing the last session of the EBP
  Providers will take an EBP knowledge and MI skills test of 25 questions from a bank of questions produced by the EBP developer.
Change In Provider Self-Efficacy for EBP Implementation | 1) prior to starting the trial (baseline) but after completing the training for the EBP and the ISS 2) within two weeks of completing the last session of the EBP
  Providers will report their self-efficacy regarding EBP implementation. Ten items from two subscales (change commitment, change efficacy) of the Readiness for Change instrument (Shea et al.) will be used to measure self-efficacy to implement the EBP.
Provider Fidelity to EBP - Component Coverage | during the 5 or 6 week EBP trial, after each session is completed
  Providers will report on their component coverage after each session during the 5 or 6 weeks of the program trial by indicating for each component whether it was fully completed, partially completed, or not completed.
Provider Fidelity to EBP - MI Quality of Delivery | during the 5 or 6 week EBP trial, after each session is completed
  Providers will report on their MI quality of delivery after each session during the 5 or 6 weeks of the program trial by completing a 10-item MI Self-Assessment questionnaire from the MIA Step Manual (NIDA/SAMHSA).
Provider Fidelity to EBP - Participant Responsiveness | during the 5 or 6 week EBP trial, after each session is completed
  Providers will report on participant responsiveness after every session during the 5 or 6 weeks of the program trial by completing a 6-item questionnaire measuring youth engagement.
Provider Perceptions of EBP - Usage Rating | within two weeks after completing the last session of the EBP
  Providers will report on their perceptions of the EBP by completing 26 items from the revised Usage Rating Profile-Intervention (URPI-R) that will measure: (a) acceptability, (b) understanding, (c) feasibility, (d) system climate, and (e) system support.
Provider Perceptions of EBP - Appropriateness | within two weeks after completing the last session of the EBP
  Providers will report on their perceptions of the EBP by completing eight items from the Training/Practice Acceptability/Feasibility/Appropriateness Scale (TPA) measuring appropriateness.
Provider Perceptions of EBP - Adoption | within two weeks after completing the last session of the EBP
  Providers will report on their EBP usage and adoption by completing the result demonstrability subscale from the Adoption of an IT innovation (AITI).
Change in Youth Beliefs, Attitudes toward Substance Use | 1) prior to starting the trial (baseline) 2) within two weeks after completing the last session of the EBP.
  Youth will report on their attitudes and beliefs toward substance use by completing questions obtained from the EBP developer. These questions will assess: (a) beliefs and attitudes, (b) perceived benefits, (c) perceived normative substance use, (d) intention to use in the future, (e) youth motivation, and (f) readiness to change.
Change in Youth Substance Use | 1) prior to starting the trial (baseline) 2) within two weeks after completing the last session of the EBP.
  Youth will report on their substance use by completing questions obtained from the EBP developer. These questions will assess: a) last 30 days use, b) negative consequences due to substance use, c) intention to use in the future, d) resistance self-efficacy, and e) coping strategies.

SECONDARY OUTCOMES:
Provider Fidelity to ISS | during training and during the 5 or 6 week EBP trial as providers use the ISS
  The system will collect usage data throughout the trial to document when and how the website and software are being used. Whenever providers access the ISS, information about that interaction will be captured. Usage statistics will be collected via a combination of HTTP access logs and session cookies to document the number of times a given webpagevideo//tool/resource is accessed.
Provider Perceptions of ISS - Usage Rating | within two weeks of completing the last session of the EBP
  Providers will report on their perceptions of the ISS by completing 26 items from the revised Usage Rating Profile-Intervention (URPI-R) that will measure: (a) acceptability, (b) understanding, (c) feasibility, (d) system climate, and (e) system support.
  Providers will report on their experiences with the ISS and their intent to use it beyond this study.
Provider Perceptions of ISS - Appropriateness | within two weeks of completing the last session of the EBP
  Providers will report on their perceptions of the ISS by completing eight items from the Training/Practice Acceptability/Feasibility/Appropriateness Scale (TPA) measuring appropriateness.
Provider Perceptions of ISS - Adoption | within two weeks after completing the last session of the EBP
  Providers will report on their ISS usage and adoption by completing the result demonstrability subscale from the Adoption of an IT innovation (AITI).
Provider Perceptions of ISS Characteristics - System Usability | within two weeks of completing the last session of the EBP
  Providers will report on the ISS characteristics by completing the Post-Study System Usability Questionnaire (PSSUQ) to assess: a) information quality, b) interface quality, and c) endorsement, and d) overall satisfaction with the ISS.
Provider Perceptions of ISS Characteristics - Components Usability | within two weeks of completing the last session of the EBP
  Providers will report on the ISS characteristics by completing the After Scenario Questionnaire (ASQ) to assess satisfaction and ease of use of each feature and component of the ISS (training resources, goal setting, fidelity, progress monitoring, implementation supports, and outcomes).
Cost Effectiveness of EBP with Centervention as the ISS | within 6-months of providers completing the last session of the FreeTalk EBP only
  To measure cost effectiveness, the brief Drug Abuse Treatment Cost Analysis Program (DATCAP) consisting of approximately 40 questions will be used to assess the cost of implementing a substance use EBP using Centervention as the ISS. Agency administrators will report via a phone interview costs associated with different aspects of traditional substance use EBP implementation at their agency.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa E DeRosier, PhD, Principal Investigator — CEO
Locations (1):
- 3C Institute, Durham, North Carolina, United States